CLINICAL TRIAL: NCT00793481
Title: Diffuse Optical Spectroscopy Measure Microvascular Changes in Metabolic Syndrome and Diabetes Mellitus in Order to Assess Cardiovascular Disease Risk.
Brief Title: Vascular Reactivity in Metabolic Syndrome and Diabetic Patients Using Diffuse Optical Spectroscopy
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Ping Wang, M.D., Professor of Medicine, University of California, Irvine
Other Study IDs: 20086415
Record Dates: First submitted 2008-11-14; First posted 2008-11-19 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus
Keywords: Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnostic tool: Diffuse Optical Spectroscopy non-invasively measure changes in the microvasculature
  Interventions: Device: Diffuse Optical Spectroscopy

INTERVENTIONS:
Device: Diffuse Optical Spectroscopy — Diffuse Optical Spectroscopy non-invasively measure changes in the microvasculature

SUMMARY:
Metabolic Syndrome is a highly prevalent condition that is comprised of several major clustering factors that increase the risk for developing cardiovascular disease. Diffuse Optical Spectroscopy is a non-invasively measure can show changes in the microvasculature of human. Diffuse Optical Spectroscopy measures the optical absorption and scattering properties of near-infrared light in tissues such as muscle in order to quantify the absolute concentration of oxygenated and deoxygenated hemoglobin, water, and lipids. It provides quantitative and functional information on the microvasculature related to tissue perfusion, metabolic changes, and indicators of tissue damage.

DETAILED DESCRIPTION:
The researchers can use Diffuse Optical Spectroscopy to monitor changes in the microvasculature of patients with Metabolic Syndrome and diabetic mellitus, and patients with Diabetic Peripheral and Autonomic Neuropathy, versus non-diseased and predisposed subjects by evaluating the changes in oxygen metabolism. The Diffuse Optical Spectroscopy measure the changes in the concentration and oxygen saturation of hemoglobin in the microvasculature under stress, for example, during exercise and in response to changes in breathing habits. The sensitivity of Diffuse Optical Spectroscopy to tissue hemodynamics provides an impressive arena of useful clinical applications..

ELIGIBILITY:
Inclusion Criteria:

* Adult ages of 45 to 75
* Have been clinically diagnosed with Type II Diabetes Mellitus
* Have a diagnosis of Metabolic Syndrome

Exclusion Criteria:

* taking light-sensitive drugs for use in photodynamic therapy
* pregnant

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic, community sample
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Changes in Microvascular | 4 weeks
  Diffuse Optical Spectroscopy non-invasively measure changes in the microvasculature

CONTACTS AND LOCATIONS:
Overall Officials: Ping H Wang, M.D., Principal Investigator — Joslin Diabetes Center,UCI; Bruce Tromberg, PhD, Study Director — Beckman Laser Institute
Locations (1):
- Beckman Laser Institute Medical clinic, Irvine, California, United States